CLINICAL TRIAL: NCT06554197
Title: Evaluation of Cytomegalovirus and Epstein-Barr Virus Specific Immune Reformulation in Prophylaxis for Cytomegalovirus in Haploid Hematopoietic Stem Cell Transplantation
Brief Title: Evaluation of CMV/EBV-CMI in Haploid HSCT
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: CMV/EBV-CMI
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cytomegalovirus Infections; Epstein-Barr Virus Infections
MeSH Terms: conditions — Cytomegalovirus Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMV/EBV-CMI — The CMV/EBV-CMI is tested before conditioning regimen and 30 days, 45 days, 60 days, 90 days, 120 days, 180 days after transplantation.

SUMMARY:
The purpose of this prospective, open-label, Single Arm, single-center study is to evaluate the cytomegalovirus and Epstein-Barr virus specific immune reestablishment for patients with hemopathy undergoingin prophylaxis for cytomegalovirus in haploid hematopoietic stem cell transplantation(haplo-HSCT) .

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed with hemopathy.
2. All patients should have the indication of Haploidentical hematopoietic stem cell transplant and receive the prophylaxis for cytomegalovirus.
3. All patients should sign an informed consent document indicating that they understand the purpose of and procedures required for the study and be willing to participate in the study.

Exclusion Criteria:

Patients with any conditions not suitable for the trial (investigators' decision).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients are diagnosed with hemopathy and should have the indication of Haploidentical hematopoietic stem cell transplant and receive the prophylaxis for cytomegalovirus.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
CMV-CMI | 6 months after transplantation
  CMV specific immune reconstitution from pre-HSCT to 180 days after HSCT
EBV-CMI | 6 months after transplantation
  EBV specific immune reconstitution from pre-HSCT to 180 days after HSCT

SECONDARY OUTCOMES:
Cumulative incidence of CMV reactivation | 1 years after transplantation
  The cumulative incidences of CMV reactivation after transplantation.
Cumulative incidences of EBV reactivation | 1 years after transplantation
  The cumulative incidences of EBV reactivation after transplantation
Overall survival (OS) | 1 years after transplantation
  Overall survival (OS) is defined as the time from randomization to death resulting from any cause.
Non-relapse mortality (NRM) | 1 years after transplantation
  Non-relapse mortality (NRM) is defined as the time from enrollment to death of any causes other than hematologic disease relapse.
Relapse-related mortality (RRM) | 1 years after transplantation
  Relapse-related mortality (RRM) is defined as the time from enrollment to death of relapse.
GVHD-free and relapse-free survival (GRFS) | 1 years after transplantation
  GRFS is defined as the time from graft infusion to the onset of grades 3 to 4 aGVHD, moderate to severe cGVHD, or relapse/disease progression/death.
Cumulative incidences of aGVHD | 100 days after transplantation
  The diagnosis and grading of aGVHD are based on the modified Glucksberg grading standard.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided